CLINICAL TRIAL: NCT03234803
Title: Metal-reinforced Flexible Poly-amide Complete Denture Versus Heat-cured Poly-methyl Methacrylate in Terms of Oral Health Related Quality of Life; Randomized Clinical Trial
Brief Title: Measuring Quality of Life of Poly-amide Complete Dentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Magdy Ibrahim, Internal resident at removable prosthodontic department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: polyamide_complete dentures
Record Dates: First submitted 2017-07-27; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Denture, Complete
MeSH Terms: interventions — Nylons; Polymethyl Methacrylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- poly-amide (Experimental): poly-amide is a thermoplastic material recently introduced to be used as a complete denture material, that provide excellent aesthetics and flexibility.
  Interventions: Other: poly-amide
- poly-methyl methacrylate (Active Comparator): poly-methyl methacrylate has been commonly used as a material for constructing complete dentures and proved to have high success rate and considered to be gold standard.
  Interventions: Other: poly-methyl methacrylate

INTERVENTIONS:
Other: poly-amide — new denture base material
  Other Names: Nylon
  Arms: poly-amide
Other: poly-methyl methacrylate — gold standard for denture base materials
  Arms: poly-methyl methacrylate

SUMMARY:
Polymethyl methacrylate have been used since 1937 as a gold standard for a denture base material because of its several advantages as; good esthetics, adequate strength, easy repair and simple processing techniques. As any material it has some problems as polymerization shrinkage, low impact and flexural properties and low fatigue resistance2. So polyamide was introduced into dentistry to be used as a denture base material in order to solve these problems. Polyamide denture base materials have some superior properties than PMMA as; High impact & flexural strength, excellent esthetics and less release of residual monomers4. Although being an advantage from the point of patient satisfaction, flexural property considered to be a contraindication for a denture base material.

The invistigators' trial is done in order to improve rigidity of a polyamide material as well as to improve oral health related quality of life in comparison to heat cured polymethyl methacrylate.

ELIGIBILITY:
Inclusion Criteria:

- i. Male or female patient with age range (45-55) and in good medical condition ii. All patients have skeletal Angle's class I maxillo-mandibular relationship and have sufficient inter-arch distance.

iii. Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.

iv. Free from any tempro-mandibular joint disorder. v. The patients have good oral hygiene.

Exclusion Criteria:

- i. Patients having hormonal disorders as diabetes, thyroid or parathyroid hormonal diseases were not included.

ii. Patient with xerostomia or excessive salivation. iii. Patient with abnormal tongue behavior and/or size. iv. No intraoral soft and hard tissue pathosis

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
oral health related quality of life | one month
  OHIP-49 questionnaire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ali IL, Yunus N, Abu-Hassan MI. Hardness, flexural strength, and flexural modulus comparisons of three differently cured denture base systems. J Prosthodont. 2008 Oct;17(7):545-9. doi: 10.1111/j.1532-849X.2008.00357.x. Epub 2008 Aug 26. PMID 18761582
- [Background] Wadachi J, Sato M, Igarashi Y. Evaluation of the rigidity of dentures made of injection-molded materials. Dent Mater J. 2013;32(3):508-11. doi: 10.4012/dmj.2013-061. PMID 23719015
- [Background] Schwindling FS, Rammelsberg P, Stober T. Effect of chemical disinfection on the surface roughness of hard denture base materials: a systematic literature review. Int J Prosthodont. 2014 May-Jun;27(3):215-25. doi: 10.11607/ijp.3759. PMID 24905261